CLINICAL TRIAL: NCT06195358
Title: Mobile Health Intervention to Promote Positive Infant Health Outcomes in Guatemala
Brief Title: Mobile Health Intervention for Infants in Guatemala (18-m Intervention)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Brigham and Women's Hospital, Boston USA (Unknown); Wuqu' Kawoq - Maya Health Alliance, Tecpán Guatemala (Unknown)
Responsible Party: Principal Investigator, Beth Smith, Associate Professor of Pediatrics (USC Faculty/Non Physician CWR), Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-21-00168_18-month; R33HD107983 (NIH)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Infant Development
Keywords: early childhood development; LMIC; Guatemala; mHealth; smartphone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): The control arm will receive printed caregiving materials.
  Interventions: Other: Printed Caregiving Materials
- Intervention Arm (Experimental): The intervention arm will receive the smartphone application.
  Interventions: Device: Mobile Health (Smartphone) Application

INTERVENTIONS:
Device: Mobile Health (Smartphone) Application — The intervention arm will receive the smartphone application, which has been designed to engage primary caregivers directly in the active monitoring of their infants' development, and to provide tailored feedback and support for the provision of nurturing care. Study staff will make an initial home visit (less than an hour) to install the application on the caregiver phone and demonstrate use and collect baseline data. Subsequently, in the intervention arm, staff will make monthly visits (approximately 15 minutes duration) to assess functionality of the smartphone and answer questions/reinforce use.
  Arms: Intervention Arm
Other: Printed Caregiving Materials — The control arm will receive printed caregiving materials. In the control arm, staff will make monthly visits (approximately 15 minutes duration) to ask if there are questions about the printed caregiving materials.
  Arms: Control Arm

SUMMARY:
Promoting optimal development for children at risk in low- and middle-income countries (LMICs) is an important global health priority. Supporting caregivers to provide nurturing care is an evidence-based strategy, however feasibility of scaling-up this supporting is limited by competing demands on health workers' time. For infant development, mHealth technologies have the potential to solve this problem by providing tailored content directly to caregivers, involving and empowering them to promote infant development, promoting and facilitating interactions with health workers when areas of concern are identified and, therefore, expanding the reach of healthcare systems. Following a pilot feasibility study, this current study will examine the effectiveness of a caregiver-directed smartphone application to directly engage first-time caregivers in rural Guatemala and support early childhood development.

DETAILED DESCRIPTION:
Rationale: According to recent estimates, nore than 40% of children under age 5 residing in low- and middle-income countries (LMICs)-250 million children in total-are at risk of not reaching their developmental potential due to living in environments with malnutrition, poverty, and lack of early stimulation. Mobile health (mHealth) technology represents an efficient strategy for scaling interventions to promote infant development.

Intervention: Individually-randomized controlled trial of mHealth application compared to paper caregiving materials. Length of intervention = 18 months.

Objectives and purpose: We will test the effectiveness of a smartphone application that will directly engage caregivers in providing nurturing care to at-risk infants. We will assess effectiveness of the mHealth application compared to paper caregiving materials by comparing group differences in Bayley scores after 18 months.

Study population: first-time parents of newborn infants, newborn infants.

ELIGIBILITY:
Inclusion Criteria:

* first-time caregivers with an infant in the eligible age range (0-4 weeks)
* infant from singleton birth
* infant from full-term (> 37 weeks gestation) birth

Exclusion Criteria:

* Presence of acute malnutrition/wasting or severe medical illness (heart disease, kidney disease, congenital abnormality) in the infant
* medical need for supplementation of breastfeeding
* caregiver not literate

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference between study arms in Composite Language Score | 18 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 47-153
Difference between study arms in Composite Motor Score | 18 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 46-154
Difference between study arms in Composite Cognitive Score | 18 months
  Using the Bayley Scales of Infant Development, 4th Edition (BSID4), higher scores better, scale range 55-145

SECONDARY OUTCOMES:
Change in the Home Observation for Measurement of the Environment Scale (HOME) Raw Score | Change from 0 to 18 months
  Raw score range 0-45, higher scores better

CONTACTS AND LOCATIONS:
Overall Officials: Beth Smith, PT, DPT, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Wuqu' Kawoq/ Maya Health Alliance, Chimaltenango, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared via NICHD DASH
Supporting Information: Study Protocol
Time Frame: data will become available upon completion of the study and publication of primary paper and will remain available indefinitely.
Access Criteria: per NICHD DASH procedures
URL: https://dash.nichd.nih.gov/